CLINICAL TRIAL: NCT01228474
Title: A Prospective, Randomized, Controlled Trial Comparing SET vs DET in an Oocyte Donation Programme
Brief Title: Single Embryo Transfer vs. Double Embryo Transfer in an Oocyte Donation Programme
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the high number of multiples pregnancies in the double embryo transfer group, we have decided to stop the enrollment of patients at 07/31/2012
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Ignacio Rodriguez, Bsc, Fundacion Dexeus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEX003
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Infertility; Oocyte Recipient; Single Embryo Transfer/Double Embryo Transfer; Cumulative Pregnancy Rate; Multiple Pregnancy
MeSH Terms: conditions — Infertility

ARMS (2):
- SET (Experimental): Single embryo transfer
  Interventions: Other: Select the Number of embryos to transfer
- DET (Active Comparator): Double embryo transfer
  Interventions: Other: Select the Number of embryos to transfer

INTERVENTIONS:
Other: Select the Number of embryos to transfer — Select the Number of embryos to transfer

SUMMARY:
Experimental study to assess the efficacy of single embryo transfer (SET) with respect to double embryo transfer (DET) in an oocyte donation programme, 160 recipients will be randomized in two groups

ELIGIBILITY:
Inclusion Criteria:

* patients under their first or second cycle of a synchronous donation
* to have a minimum of 5 available embryos to transfer
* patients who accept transfers of frozen-thawed embryos

Exclusion Criteria:

* medical indications to transfer only one embryo (Turner Syndrome, uterine surgical history, uterine myomas,…)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Cumulative pregnancy rate | at 12 months of fresh embryo transfer (time considered enough in order to do a minimum of one frozen-thawed cycle if pregnancy is not achieved with the fresh cycle

SECONDARY OUTCOMES:
Cumulative live birth rate
Multiple pregnancy rate
Time needed to achieve the pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Departamento de Obstetricia, Ginecología y Reproducción. Institut Universitari Dexeus, Barcelona, Barcelona, Spain

REFERENCES:
- [Background] Soderstrom-Anttila V, Vilska S. Five years of single embryo transfer with anonymous and non-anonymous oocyte donation. Reprod Biomed Online. 2007 Oct;15(4):428-33. doi: 10.1016/s1472-6483(10)60369-0. PMID 17908406
- [Background] Soderstrom-Anttila V, Vilska S, Makinen S, Foudila T, Suikkari AM. Elective single embryo transfer yields good delivery rates in oocyte donation. Hum Reprod. 2003 Sep;18(9):1858-63. doi: 10.1093/humrep/deg384. PMID 12923139
- See also: Related Info — http://www.dexeus.com